CLINICAL TRIAL: NCT07339761
Title: SPICE: Supporting Sexual Health in Bladder Cancer Patients: A Sequential Mixed-Methods Intervention Study
Brief Title: Supporting Sexual Health in Bladder Cancer Patients: A Sequential Mixed-Methods Intervention Study
Acronym: SPICE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: DUAUHSPICE
Record Dates: First submitted 2025-12-10; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Bladder Cancer; Non-Muscle-Invasive Bladder Cancer (NMIBC); Muscle-Invasive Bladder Carcinoma
Keywords: Sexual Health; Bladder Cancer; Sexual Rehabilitation
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: * Study 1a (Development phase): A qualitative, exploratory study to develop a sexological intervention with patient and clinician involvement.
  * Study 1b (Feasibility phase): A one-armed feasibility trial assessing the implementation and acceptability of the intervention among patients with muscle-invasive bladder cancer (MIBC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (study 1b) (Experimental)
  Interventions: Other: Sexological Support

INTERVENTIONS:
Other: Sexological Support — Results from Study 1a will inform the development and refinement of the intervention to be tested in the feasibility phase (Study 1b).

SUMMARY:
Despite increasing recognition of sexual dysfunction and sexual distress as important survivorship issues in oncology, research and clinical attention remain uneven across cancer types. This imbalance is particularly evident in bladder cancer, where sexual health has received limited research and clinical attention. However, existing studies demonstrate substantial sexual dysfunction and reduced intimacy among patients following disease and treatment.

The treatment of bladder cancer is a multimodal and multidisciplinary discipline. Low-risk non-muscle-invasive bladder cancer (NMIBC) is treated by transurethral resection of the bladder (TURB) alone, while recurrent intermediate- and high-risk NMIBC undergo a combination of TURB and adjuvant intravesical instillation therapy. For patients with muscle-invasive bladder cancer (MIBC) and specific high-risk NMIBC cases, the first-line treatment option is radical cystectomy with urinary diversion, with or without neoadjuvant chemotherapy.

These treatment modalities are known to have a negative impact on sexual function, and studies in both men and women demonstrate profound impairments in sexual function, intimacy, and body image after treatment. Among men, erectile and ejaculatory dysfunction are prevalent for this patient group and frequently associated with diminished sexual satisfaction and body-image concerns. Likewise, women experience loss of sexual desire, orgasmic disorders, dyspareunia, and vaginal dryness following cystectomy.

A targeted literature search further identified no contemporary sexology-focused interventional or feasibility trials specifically in bladder cancer (neither MIBC or NMIBC). Existing evidence on the topic is largely descriptive or addresses non-sexological rehabilitation, demonstrating a evidence gap[1].

Qualitative research has also explored informational and psychosocial needs among bladder cancer patients, revealing limited communication about sexual health and unmet needs for professional support. Such studies provide valuable insight into patient experiences but have not yet translated this knowledge into the development of structured, sexological interventions.

Evidence from other cancer populations demonstrates that counselling and psychoeducational programmes addressing intimacy and sexuality are both feasible and beneficial, suggesting that similar interventions could be adapted for bladder cancer care.

To develop a relevant and acceptable intervention, it is essential to understand how patients themselves perceive their sexual health challenges, informational needs, and preferences for professional support regarding sexual health.

This project therefore consists of two sequential sub-studies:

* Study 1a (Development phase): A qualitative, exploratory study to develop a sexological intervention with patient and clinician involvement.
* Study 1b (Feasibility phase): A one-armed feasibility trial assessing the implementation and acceptability of the intervention among patients with muscle-invasive bladder cancer (MIBC).

ELIGIBILITY:
Inclusion Criteria study 1a:

* The participant has one of the following diagnoses and received initial treatment approximately 12 months ago:

  1. Non-muscle-invasive bladder cancer treated with transurethral resection of the bladder (TUR-B)
  2. Non-muscle-invasive bladder cancer treated with TUR-B and subsequent intravesical instillation therapy with chemotherapy or immunotherapy
  3. Muscle-invasive bladder cancer treated with cystectomy (removal of the bladder)
* The participant has experienced changes and/or difficulties in sexual function related to the cancer diagnosis and/or its treatment
* The participant speaks and understands Danish
* The participant is aged 18 years or older
* The participant has read and understood the oral and written study information
* The participant has provided written informed consent

Exclusion Criteria study 1a:

* The participant has a history of other cancers located in the pelvic region, including rectal cancer, sarcomas, uterine cancer, cervical cancer, ovarian cancer, prostate cancer, or penile cancer
* The participant has a history of breast cancer

Inclusion Criteria study 1b:

* The participant is diagnosed with Muscle-invasive bladder cancer treated with cystectomy (removal of the bladder)
* The participant speaks and understands Danish
* The participant is aged 18 years or older
* The participant has read and understood the oral and written study information
* The participant has provided written informed consent

Exclusion Criteria study 1b:

* The participant has a history of other cancers located in the pelvic region, including rectal cancer, sarcomas, uterine cancer, cervical cancer, ovarian cancer, prostate cancer, or penile cancer
* The participant has a history of breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Study 1a: Patient-perceived sexual health challenges identified through semi-structured qualitative interviews | 1 year
  Patient perceptions of sexual health challenges will be explored through semi-structured individual interviews. Interviews will be audio-recorded, transcribed verbatim, and analyzed using thematic analysis. Results will be reported as descriptive themes representing common challenges across participants.
Study 1a: Patient informational needs regarding sexual health identified through semi-structured qualitative interviews | 1 year
  Patient informational needs related to sexual health will be assessed through semi-structured individual interviews. Interview transcripts will be analyzed using thematic analysis, and results will be reported as themes describing shared informational needs.
Study 1a: Patient preferences for professional sexual health support identified through semi-structured qualitative interviews | 1 year
  Patient preferences for professional sexual health support will be explored using semi-structured individual interviews. Data will be analyzed using thematic analysis, and findings will be reported as themes describing preferred type, timing, and format of support.
Study 1b: Recruitment rate | 2 years
  Recruitment rate will be defined as the number of participants enrolled divided by the number of eligible participants approached during the recruitment period.
Study 1b: Retention rate | 2 years
  Retention rate will be defined as the proportion of enrolled participants who complete all required study assessments.
Study 1b: Adherence to study protocol | 2 years
  Protocol adherence will be assessed as the proportion of participants who complete the intervention according to the predefined study procedures.
Study 1b: Response rate to patient-reported outcome measures | 2 years
  Response rate will be defined as the proportion of completed patient-reported outcome questionnaires out of the total number of questionnaires distributed.
Study 1b: Data completeness of patient-reported outcome measures | 2 years
  Data completeness will be assessed as the proportion of fully completed items across all patient-reported outcome measures.

SECONDARY OUTCOMES:
Study 1b: Sexual function assessed by the Female Sexual Function Index (FSFI) | 2 years
  Sexual function will be assessed using the Female Sexual Function Index (FSFI). The total score ranges from 2 to 36, with higher scores indicating better sexual function.
Study 1b: Sexual distress assessed by the Female Sexual Distress Scale-Revised (FSDS-R) | 2 years
  Sexual distress will be measured using the Female Sexual Distress Scale-Revised (FSDS-R). Total scores range from 0 to 52, with higher scores indicating greater sexual distress.
Study 1b: Wellbeing assessed by the WHO-5 Well-Being Index | 2 years
  Wellbeing will be assessed using the WHO-5 Well-Being Index. Scores range from 0 to 100, with higher scores indicating better wellbeing.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Aarhus University Hospital, Aarhus, Denmark